CLINICAL TRIAL: NCT01108419
Title: Evaluation of the Safety and Tolerance of a New Fermented Food in Healthy Adults
Brief Title: Evaluation of Dose-effect of a New Fermented Food in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NU327
Record Dates: First submitted 2010-03-29; First posted 2010-04-22 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: healthy adults
MeSH Terms: interventions — Cultured Milk Products

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 = Test Product normal dose (Active Comparator): Fermented dairy product containing probiotics - normal dose
  Interventions: Other: Fermented dairy product
- 2 = Test Product high dose (Active Comparator): Fermented dairy product containing probiotics - high dose
  Interventions: Other: Fermented dairy product
- 3 = Control Product normal dose (Sham Comparator): Non-fermented dairy product - normal dose
  Interventions: Other: milk-based non-fermented dairy product
- 4 = Control Product high dose (Sham Comparator): Non-fermented dairy product - high dose
  Interventions: Other: milk-based non-fermented dairy product

INTERVENTIONS:
Other: Fermented dairy product
  Arms: 1 = Test Product normal dose; 2 = Test Product high dose
Other: milk-based non-fermented dairy product
  Arms: 3 = Control Product normal dose; 4 = Control Product high dose

SUMMARY:
The aim of the study is to assess the safety and tolerance of a new fermented food versus a control product in healthy adults during the 4-week consumption period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects after receiving a full description of the study, provide written informed consent to take part in the study.
* Free-living subject, as evaluated during the clinical examination.
* Male/female subjects aged between 18 to 55 years (bounds included).
* Subjects with a body mass index (BMI) between 18.5 ≤ BMI < 30kg/m².
* Healthy subjects (as determined by a medical examination)

Exclusion Criteria:

* Subjects with any allergy (food, respiratory…).
* Subjects that have had any surgery or intervention requiring general anaesthesia in the last 4 weeks.
* Subjects with a history of chronic metabolic or gastrointestinal disease with the exception of appendectomy.
* Subjects with chronic or iatrogenic immunodeficiency (e.g. Chemotherapy, HIV).
* Subjects presenting a severe evolutive or chronic pathology (e.g. cancer,tuberculosis, Crohn's disease, cirrhosis, multiple sclerosis, Type I diabetes…).
* Subject with eating disorders.
* Subjects with cardiac, respiratory (including asthma) or renal insufficiency, cardiomyopathy, valvulopathy and medical history of rheumatic fever.
* Subjects with special medicated diet (for obesity, anorexia, metabolic pathology…).
* For female subjects: pregnancy, breast-feeding or not willing to use/not using an acceptable method of contraception
* Subject, in the Investigator's opinion, should not be randomised.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Effect of 1 bottle/day of test versus control product on adverse events. | During the 4-week period of product consumption.
  Number of Adverse events, number of AE related to product, number of emergent AE, number of mild/moderate and severe AE, number of serious AE.
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week period of product consumption.
  Systolic/diastolic blood pressure (mmHg).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week period of product consumption.
  Heart rate (bpm).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week period of product consumption.
  Weight (kg).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week period of product consumption.
  Body mass index (kg/m²).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week period of product consumption.
  Temperature (°C).
Effect of 1 bottle/day of test versus control product on hematology. | During the 4-week period of product consumption.
  Hemoglobin (mmol/L).
Effect of 1 bottle/day of test versus control product on hematology. | During the 4-week period of product consumption.
  Hematocrit (L/L).
Effect of 1 bottle/day of test versus control product on hematology. | During the 4-week period of product consumption.
  Red blood cell, white blood cell, platelets (count/L).
Effect of 1 bottle/day of test versus control product on glucose and lipids metabolism. | During the 4-week period of product consumption.
  blood glucose (mmol/L), lipids [total cholesterol, HDL, LDL, triglycerides] (mmol/L).
Effect of 1 bottle/day of test versus control product on liver function. | During the 4-week period of product consumption.
  Blood alanine aminotransferase, aspartate aminotransferase, gamma-glutamyltransferase (IU/L).
Effect of 1 bottle/day of test versus control product on kidney function. | During the 4-week period of product consumption.
  Blood creatinin (μmol/L).
Effect of 1 bottle/day of test versus control product on thyroid function. | During the 4-week period of product consumption.
  Blood thyroid stimulating hormone (mU/L).
Effect of 1 bottle/day of test versus control product on blood marker of inflammation. | During the 4-week period of product consumption.
  Blood C-reactive protein (mmol/L)
Effect of 1 bottle/day of test versus control product on fecal marker of inflammation. | During the 4-week period of product consumption.
  Fecal calprotectin (μg/g)
Effect of 1 bottle/day of test versus control product on bowel habits. | During the 4-week period of product consumption.
  Stool frequency and consistency (Bristol Stool Scale from 1 [hard stools] to 7 [watery stools]).
Effect of 1 bottle/day of test versus control product on digestive symptoms. | During the 4-week period of product consumption.
  Frequency of abdominal pain/discomfort, abdominal bloating, flatulence, borborygmi/rumbling.

SECONDARY OUTCOMES:
Effect of 1 bottle/day of test versus control product on adverse events. | During the 4-week follow-up period and the 8-week entire study period.
  Number of Adverse events, number of AE related to product, number of emergent AE, number of mild/moderate and severe AE, number of serious AE.
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week follow-up period and the 8-week entire study period.
  Systolic/diastolic blood pressure (mmHg).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week follow-up period and the 8-week entire study period.
  Heart rate (bpm).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week follow-up period and the 8-week entire study period.
  Weight (kg).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week follow-up period and the 8-week entire study period.
  Body mass index (kg/m²).
Effect of 1 bottle/day of test versus control product vital signs. | During the 4-week follow-up period and the 8-week entire study period.
  Temperature (°C).
Effect of 1 bottle/day of test versus control product on hematology. | During the 4-week follow-up period and the 8-week entire study period.
  Hemoglobin (mmol/L).
Effect of 1 bottle/day of test versus control product on hematology. | During the 4-week follow-up period and the 8-week entire study period.
  Hematocrit (L/L).
Effect of 1 bottle/day of test versus control product on hematology. | During the 4-week follow-up period and the 8-week entire study period.
  Red blood cell, white blood cell, platelets (count/L).
Effect of 1 bottle/day of test versus control product on glucose and lipids metabolism. | During the 4-week follow-up period and the 8-week entire study period.
  blood glucose (mmol/L), lipids [total cholesterol, HDL, LDL, triglycerides] (mmol/L).
Effect of 1 bottle/day of test versus control product on liver function. | During the 4-week follow-up period and the 8-week entire study period.
  Blood alanine aminotransferase, aspartate aminotransferase, gamma-glutamyltransferase (IU/L).
Effect of 1 bottle/day of test versus control product on kidney function. | During the 4-week follow-up period and the 8-week entire study period.
  Blood creatinin (μmol/L).
Effect of 1 bottle/day of test versus control product on thyroid function. | During the 4-week follow-up period and the 8-week entire study period.
  Blood thyroid stimulating hormone (mU/L).
Effect of 1 bottle/day of test versus control product on blood marker of inflammation. | During the 4-week follow-up period and the 8-week entire study period.
  Blood C-reactive protein (mmol/L)
Effect of 1 bottle/day of test versus control product on fecal marker of inflammation. | During the 4-week follow-up period and the 8-week entire study period.
  Fecal calprotectin (μg/g)
Effect of 1 bottle/day of test versus control product on bowel habits. | During the 4-week follow-up period and the 8-week entire study period.
  Stool frequency and consistency (Bristol Stool Scale from 1 [hard stools] to 7 [watery stools]).
Effect of 1 bottle/day of test versus control product on digestive symptoms. | During the 4-week follow-up period and the 8-week entire study period.
  Frequency of abdominal pain/discomfort, abdominal bloating, flatulence, borborygmi/rumbling.
Effect of 3 bottles/day of test versus control product on adverse events. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Number of Adverse events, number of AE related to product, number of emergent AE, number of mild/moderate and severe AE, number of serious AE.
Effect of 3 bottles/day of test versus control product vital signs. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Systolic/diastolic blood pressure (mmHg).
Effect of 3 bottles/day of test versus control product vital signs. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Heart rate (bpm).
Effect of 3 bottles/day of test versus control product vital signs. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Weight (kg).
Effect of 3 bottles/day of test versus control product vital signs. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Body mass index (kg/m²).
Effect of 3 bottles/day of test versus control product vital signs. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Temperature (°C).
Effect of 3 bottles/day of test versus control product on hematology. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Hemoglobin (mmol/L).
Effect of 3 bottles/day of test versus control product on hematology. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Hematocrit (L/L).
Effect of 3 bottles/day of test versus control product on hematology. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Red blood cell, white blood cell, platelets (count/L).
Effect of 3 bottles/day of test versus control product on glucose and lipids metabolism. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  blood glucose (mmol/L), lipids [total cholesterol, HDL, LDL, triglycerides] (mmol/L).
Effect of 3 bottles/day of test versus control product on liver function. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Blood alanine aminotransferase, aspartate aminotransferase, gamma-glutamyltransferase (IU/L).
Effect of 3 bottles/day of test versus control product on kidney function. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Blood creatinin (μmol/L).
Effect of 3 bottles/day of test versus control product on thyroid function. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Blood thyroid stimulating hormone (mU/L).
Effect of 3 bottles/day of test versus control product on blood marker of inflammation. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Blood C-reactive protein (mmol/L)
Effect of 3 bottles/day of test versus control product on fecal marker of inflammation. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Fecal calprotectin (μg/g)
Effect of 3 bottles/day of test versus control product on bowel habits. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Stool frequency and consistency (Bristol Stool Scale from 1 [hard stools] to 7 [watery stools]).
Effect of 3 bottles/day of test versus control product on digestive symptoms. | During the 4-week period of product consumption, the 4-week follow-up period and the 8-week entire study period.
  Frequency of abdominal pain/discomfort, abdominal bloating, flatulence, borborygmi/rumbling.
Effect of 1 bottle/day of test versus control product on test product strains detection and quantification in feces. | During the 4-week period of product consumption and after 4-week follow-up period.
  Concentration of test product bacterial strains in feces by quantitative PCR (bacterial cells/g of feces).
Effect of 1 bottle/day of test versus control product on microbiota analysis in feces. | During the 4-week period of product consumption and after 4-week follow-up period.
  Gut microbiota analysis by sequencing approaches (16S rRNA and shotgun sequencing): Alpha (index) and beta-diversity (distance).
Effect of 1 bottle/day of test versus control product on microbiota analysis in feces. | During the 4-week period of product consumption and after 4-week follow-up period.
  Gut microbiota analysis by sequencing approaches (16S rRNA and shotgun sequencing): relative abundance of bacterial genera (%) and metabolic pathways (%).
Effect of 3 bottles/day of test versus control product on test product strains detection and quantification in feces. | During the 4-week period of product consumption and after 4-week follow-up period.
  Concentration of test product bacterial strains in feces by quantitative PCR (bacterial cells/g of feces).
Effect of 3 bottles/day of test versus control product on microbiota analysis in feces. | During the 4-week period of product consumption and after 4-week follow-up period.
  Gut microbiota analysis by sequencing approaches (16S rRNA and shotgun sequencing): Alpha (index) and beta-diversity (distance).
Effect of 3 bottles/day of test versus control product on microbiota analysis in feces. | During the 4-week period of product consumption and after 4-week follow-up period.
  Gut microbiota analysis by sequencing approaches (16S rRNA and shotgun sequencing): relative abundance of bacterial genera (%) and metabolic pathways (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Harrison Clinical Research Clinical Unit, Hilblestrasse 54, München, Germany